CLINICAL TRIAL: NCT07022964
Title: A Multicenter, Open-Label, Non-Randomized, Single-Arm Phase I/II Clinical Study of Autologous and New Donor CD7 CAR-T Cells for Relapsed or Refractory Mature T-Cell Lymphomas
Brief Title: CD5 CAR T-Cell Therapy for r/r T-cell Lymphomas
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Collaborators: Ruijin Hospital (Other); Shanghai Liquan Hospital (Other)
Responsible Party: Principal Investigator, Jing Pan, Director of Dept of Hemato-Oncology and Immunotherapy, Beijing GoBroad Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJGBYY-IIT-LCYJ-2025-032
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: T-Cell Non-Hodgkin Lymphoma; T-cell Lymphoma (PTCL and CTCL)
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD5 CAR-T therapy (Experimental): Enrolled patients were treated with anti-CD7 CAR-T cells, with or without allo-HSCT bridging.
  Interventions: Drug: CD5 CAR-T cells infusion

INTERVENTIONS:
Drug: CD5 CAR-T cells infusion — Approximately 3-5 days prior to CD5 CAR-T cell infusion, subjects are treated with FC regimen (fludarabine and cyclophosphamide) for lymphodepletion. CAR-T cell infusion are performed 48 h after completion of chemotherapy.

SUMMARY:
This is a multi-center, open-label, non-randomized, single-arm clinical trial. Refractory/relapse T-NHL patients are treated with autologous and allogeneic CD5 CAR T-cell therapy. The primary objective is to prospectively evaluate the safety of CD5 CAR T cell bridging to HSCT in the treatment of r/r T-NHL. The primary endpoint is the type and incidence of dose limiting toxicity (DLT) within 21 days after CD5 CAR-T cell infusion. A total of 36 subjects is estimated to be enrolled.

ELIGIBILITY:
Inclusion Criteria (Patients who met all the inclusion criteria were eligible for enrolment):

* Relapsed or refractory CD7-positive T-cell lymphomas that were treated with with standard chemotherapy, with poor prognosis from currently available treatments at and no available treatment options (e.g., HSCT or chemotherapy);
* Male or female, age 14-70;
* Eastern Cooperative Oncology Group (ECOG) Physical Status Score 0-2;
* life expectancy is at least 60 days;
* Subjects should be capable of understanding and signing the informed consent form prior to any screening procedures. Subjects are willing to follow the study visit schedule and associated study procedures as specified in the protocol. Candidates between the ages of 19-70 years old will need to be sufficiently aware of and capable of signing the informed consent form; underage candidates between the ages of 14-18 years old will need to be sufficiently aware of the informed consent form and their legal guardian will also need to sign the informed consent form separately.

Exclusion Criteria (Patients who fulfil any of the following criteria may not be enrolled):

* Patients with history of allogeneic HSCT but PBMNC is not available from prior- transplant donor for preparation of CAR T cells and peripheral blood tumour load >30%; patients without history of allogeneic HSCT and peripheral blood tumour load >30%;
* Intracranial hypertension or cerebral impaired consciousness;
* Symptomatic heart failure or severe arrhythmia;
* Symptoms of severe respiratory failure;
* With other types of malignancy;
* Diffuse intravascular coagulation;
* Serum creatinine and/or urea nitrogen ≥ 1.5 times the normal value;
* With sepsis or other uncontrollable infection;
* Suffering from uncontrollable diabetes mellitus;
* Severe mental disorders;
* Have significant intracranial lesions on cranial MRI;
* Organ transplantation (excluding haematopoietic stem cell transplantation) history;
* Female patients (patients of childbearing potential) with positive blood HCG test;
* Hepatitis (including hepatitis B and C) and positive screening for AIDS and syphilis.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 21 days
  Incidence and type of dose-limiting toxicity(DLT) within 21 days of CD7 CAR-T infusion.
Adverse events (AEs) | 21 days
  Total number, incidence and severity of adverse events (AEs) within 21 days of CD7 CAR-T infusion.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 21, 90 days
  The assessment of ORR by dose group at 21 and 90 Days after CD7 CAR T infusion.
Duration of response (DOR) | up to 2 years
  DOR is defined as the date when CR response criteria are first met to the date of relapse or death caused by T-NHL in the absence of documented relapse

CONTACTS AND LOCATIONS:
Overall Officials: Tengyu Wang, Ph.D, Principal Investigator — Beijing GoBroad Hospital, Beijing, Beijing 102200
Locations (3):
- China (3):
  - Beijing GoBroad Hospital, Beijing
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Liquan Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided